CLINICAL TRIAL: NCT02252614
Title: Efficacy of Intravenous Naproksen Sodium+Codein and Paracetamol+Codein on Postoperative Pain and Contramal Consumption After a Lumbar Disk Surgery
Brief Title: Efficacy of Intravenous Naproksen Sodium+Codein and Paracetamol+Codein on Postoperative Pain on Postoperative Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Reyhan Polat, Medical Doctor, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DiskapiYBERH
Record Dates: First submitted 2014-09-26; First posted 2014-09-30 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Postoperative Pain, PCA Contramal Consumption
Keywords: naproxen sodium+codein, paracetamol+codein,lumbar disc surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Naproxen sodium codein (Active Comparator): Preoperative Naproxen sodium codein administered, pain intensity measured by the visual analogue scale, and contramal consumption and related side effects evaluated.
  Interventions: Drug: naproxen sodium codein
- Paracetamol codein (Experimental): Preoperative paracetamol codein administrered, pain intensity measured by the visual analogue scale, and contramal consumption and related side effects evaluated.
  Interventions: Drug: paracetamol codein
- Placebo tablet (Placebo Comparator): Preoperative placebo tablet administered, pain intensity measured by the visual analogue scale, and contramal consumption and related side effects evaluated.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: naproxen sodium codein — Pain intensity, contramal consumption
  Other Names: Apranax plus
  Arms: Naproxen sodium codein
Drug: paracetamol codein — Pain intensity, contramal consumption
  Other Names: Geralgine K tablet
  Arms: Paracetamol codein
Drug: Placebo — Pain intensity, contramal consumption
  Other Names: Placebo tablet
  Arms: Placebo tablet

SUMMARY:
Comparition the analgesic effects of intravenous naproksen sodyum+codein with that of paracetamol+codein on postoperative pain and contramal consumption during the first 24 hour after a lumbar disk surgery.

DETAILED DESCRIPTION:
Patients were treated using patient-controlled analgesia with contramal for 24 hours after a lumbar disk surgery and randomized to receive IV naproksen sodium+codein, paracetamol+codein or isotonic saline (placebo).

The primary endpoint was pain intensity measured by the visual analogue scale, and secondary endpoints were contramal consumption and related side effects.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists 1 or 2 status patients scheduled for elective lumbar disk surgery under general anesthesia

Exclusion Criteria:

* Patients, known allergies to any of the drugs used in this study
* eptic ulcer disease, hepatic and renal dysfunction, emergency surgery, or inability to provide informed consent (eg, mental disorders)

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2014-09; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity, contramal consumption | Postoperative 24 hour

SECONDARY OUTCOMES:
side effects, nausa, vomiting | postoperative 24 hour

CONTACTS AND LOCATIONS:
Overall Officials: Reyhan Polat, MD, Principal Investigator — Diskapi YBERH